CLINICAL TRIAL: NCT02288455
Title: A Prospective, Non-Randomized, Multi-Center Clinical Investigation of the Safety and PeRformancE of GT UroLogIcal, LLC's ArtiFicial Urinary Sphincter (RELIEF II)
Brief Title: Clinical Investigation of GT UrologIcal, LLC's Artificial Urinary Sphincter (RELIEF II)
Acronym: RELIEFII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GT Urological, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP13-101
Record Dates: First submitted 2014-11-06; First posted 2014-11-11 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Male Stress Urinary Incontinence
Keywords: SUI, incontinence, sphincter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RELIEF II - GTU AUS (Experimental): Prospective, non-randomized multi-center study testing the safety and efficacy of the GTU Artificial Urinary Sphincter device in males with stress urinary incontinence.
  Interventions: Device: GTU Artificial Urinary Sphincter

INTERVENTIONS:
Device: GTU Artificial Urinary Sphincter — A totally implantable Artificial Urinary Sphincter (AUS) for the treatment of male Stress Urinary Incontinence (SUI)

SUMMARY:
The purpose of this investigation is to demonstrate the safety and efficacy of the GTU artificial urinary sphincter device in restoring continence in males who have confirmed urinary stress incontinence for a minimum of 12 months with primary etiology being radical prostatectomy or transurethral resection of the prostate (TURP).

DETAILED DESCRIPTION:
Prospective, non-randomized multi-center study testing the safety and efficacy of the GTU artificial urinary sphincter device in males with urinary incontinence.

Up to 20 sites in Europe, Australia & New Zealand

A sample size of 73 subjects is estimated to provide 80% power for efficacy. Accounting for 10% attrition, 82 subjects will be enrolled to provide non-missing data on 73 subjects.

First Subject Enrolment: July 2014 Last Subject Enrolment: September 2015 Last Subject Follow-up: September 2016 Study Primary Endpoint Completion: January 2016

Each subject will be followed for approximately 14 months. Study duration is approximately 27 months.

Subjects will be evaluated at the screening, pre-implant, implant, 6 weeks post implant for device activation, 1-month, 2-month, 3-month, 6-month, and 12-month post device activation.

The Sponsor (GT Urological, LLC) will work with a Contract Research Organization (CRO) to assist in investigative site monitoring for this clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Males > 21 years
2. Willing/able to sign informed consent
3. Has undergone radical prostatectomy or transurethral resection of the prostate or other prostate surgery prior to 6 months of the time of enrollment
4. Primary stress urinary incontinence confirmed urodynamically as dominant form of UI
5. Failed conservative incontinence treatment (see list below) for at least 6 months

   1. Pelvic exercises and bladder training
   2. Drug Therapy
   3. Biofeedback
   4. Electrical stimulation
   5. Behavioral therapy
6. Subject has severe urinary incontinence defined by:

   a. One 24-hour pad weight test ≥300 gm
7. Max urethral closure pressure < 30 cm H2O
8. Bladder capacity > 250 ml
9. Post void residual urine < 50 ml
10. Abnormal/poor compliance bladder defined by <30-40cm H2O.
11. Willing/able to comply with follow-up activities
12. Is an appropriate surgical candidate as determined by the investigator
13. Negative urine culture prior to surgery
14. Cognitive/manual capability to operate device

Exclusion Criteria:

1. Subjects considered to be vulnerable
2. Refuses or unable to sign the informed consent
3. Cannot comply with study requirements, follow-up visits and tests
4. Currently enrolled or plans to enroll in another investigational device or drug clinical trial or has completed an investigational study within 2 weeks
5. Estimated life span < 5 years
6. Recent or planned surgeries within 3 months before or 12 weeks after the implant procedure
7. Primary urge incontinence, mixed incontinence with a predominant urgency component, or urinary incontinence due to or complicated by bladder outlet obstruction
8. Has had implantation of artificial urinary sphincter prosthesis, sling, or other urogenital implant
9. Has had ProACT device explanted and the urethra is compromised as assessed by the investigator
10. Demonstrated bladder outlet obstruction (BOO) as measured by the pressure flow cystometry
11. Neurogenic bladder dysfunction not treatable/controllable by pharmacological or alternative methods
12. Uncontrolled diabetes mellitus defined as persistent blood sugar level recordings of >12mmol/l (216. mg/dl) and a glycosylated hemoglobin (HbA1C) of >9% (75mmol/mol) over the preceding 3 months
13. Active abscess or infection
14. Bladder neck or urethral stricture disease requiring > 2 regular instrumentation or dilation proximal to or at the level of the urethral sheath
15. Bladder cancer or transitional cell carcinoma requiring regular cystoscopy and/or rapidly progressive prostatic or testicular cancer
16. Needs self-intermittent catheterization
17. Diagnosed disease precluding subject from being able to recall or summarize urinary status
18. Diagnosed disease or medical condition (e.g., Parkinson's) precluding subject from being physically capable of manipulating the device
19. History of bleeding diathesis or cannot stop usage of an anti-coagulant until the International Normalized Ratio (INR) is below 1.5 or quick value >70
20. Uses an indwelling catheter or condom catheter for treatment of incontinence and is not willing to discontinue use for study assessments
21. Abnormal Prostate Screening Antigen (PSA), according to site's laboratory standards, unless further investigation confirms no signs of local recurrence
22. Known allergy to device material
23. Active or recurrent urinary tract infections (UTIs) . Recurrent defined as > 4 times over the past year
24. Urodynamic testing shows significant incontinence caused by factors other than stress incontinence
25. No anatomic abnormalities of the urethra, scrotum or penis judged to prevent implantation

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-10; Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: Improvement in pad weight defined as at least 60% improvement in pad weight from baseline to 3-months post device activation as measured by the 24-hour pad weight tests. | 3 months
  The primary efficacy endpoint is improvement in pad weight defined as at least 60% improvement in pad weight from baseline to 3-months post device activation as measured by the 24-hour pad weight tests.

SECONDARY OUTCOMES:
1-Hour Pad Weight | 3 months
  Improvement in 1- hour pad weight test results from baseline to 3-month post-device activation visit.
Pad Usage | 3 months
  Improvement in number of pads used per day from baseline to 3-month post-device activation as measured by a 3-day voiding diary.
Quality of Life Assessment | 3 months
  Improvement in Quality of Life assessments as measured by:
  * Incontinence Quality of Life (IQOL)
  * International Consultation on Incontinence Questionnaire - Male Lower Urinary Tract Symptoms (ICIQ-MLUTS)
Secondary Safety Endpoint: Summary of all adverse events | 3 months
  Summary of all adverse events
Primary Safety Endpoint | 3 months
  The primary safety endpoint is a composite of the following major device-related adverse events and/or outcomes at 3 months post-device activation as reported by the investigational site. The components of this composite safety endpoint are:
  * Infection
  * Erosion
  * Urethral atrophy
  * Device reposition
  * Device revision
  * Device removal

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Haillot, Study Director — Hôpitaux de Tours
Locations (6):
- Australia (3):
  - Urology Centre, Port Macquarie, New South Wales
  - South Coast Urology, Wollongong, New South Wales
  - St George Hospital, Sydney
- Czechia (2):
  - nemocnice Ostrava, Ostrava
  - Fakultni Thomayerova nemocnice, Prague
- Tauranga Urology Research Limited, Tauranga, New Zealand